CLINICAL TRIAL: NCT02940431
Title: Active Games: Increasing the Attractiveness of Active Video Game Play for Youth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: USDA Grand Forks Human Nutrition Research Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Other
Other Study IDs: GFHNRC406
Record Dates: First submitted 2016-10-19; First posted 2016-10-20 (Estimated); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Child; Overweight; Sedentary Lifestyle
MeSH Terms: conditions — Overweight; Sedentary Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- High Autonomy (Experimental): Children will choose active video games for use during the study.
  Interventions: Other: High Autonomy
- Low Autonomy (Experimental): Children will be assigned active video games for use during the study.
  Interventions: Other: Low Autonomy

INTERVENTIONS:
Other: High Autonomy — Children will be given two active video games (AVGs) of their choice. After two weeks, a researcher will monitor progress and exchange the AVGs and sedentary games. At each exchange, children will be allowed to select their next game.
  Arms: High Autonomy
Other: Low Autonomy — Children will be given their most-liked active video game (AVG) from the baseline relative reinforcing value assessment. After two weeks, a researcher will monitor progress and exchange the AVGs and sedentary games. At each exchange, children will receive a pre-determined game.
  Arms: Low Autonomy

SUMMARY:
The purpose of this study is to look at the effects of active video game play on youth physical activity.

DETAILED DESCRIPTION:
Child obesity is increasing worldwide and has major implications for health, both during youth and later in life. Physical activity declines sharply during adolescence, making ages 8-12 a critical period to encourage healthy exercise habits. Increased childhood weight has been linked to sedentary leisure time activities, such as video games. "Active video games" (AVGs) are now being studied as a method to increase children's interest and participation in physical activity. Although research indicates that AVG play may lead to energy expenditure comparable to light/ moderate physical activity, children prefer sedentary video games to AVGs and often find AVGs boring. Children do not play AVGs as often or with the same intensity as traditional games/sports and lose interest in them; efforts must be made to increase the appeal of AVGs so they are competitive with sedentary video games. This study will examine whether children's motivation to engage in AVG play may be increased with greater autonomy, as well as whether increasing children's motivation to play AVGs also increases their motivation to play sedentary video games.

ELIGIBILITY:
Inclusion Criteria:

* Sedentary lifestyle
* BMI between 5th and 95th percentile

Exclusion Criteria:

* taking any medications that affect energy use or eating
* actively trying to lose weight
* has any medical conditions that prevent him/her from safely joining in physical activity
* exercises more than three times per week for one hour at a time
* does not engage in more than 14 hours per week of screen-based activities
* does not own an active video game system
* plays active video games more than 30 minutes per week

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 49 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2018-05-04 (Actual); Study Completion 2018-05-04 (Actual)

PRIMARY OUTCOMES:
Change in relative reinforcing value (RRV) of active video games | Week 0, Week 6, Week 10
  RRV of active video games will be assessed by evaluating the number of responses (mouse button presses) a participant is willing to complete to gain access to active video game play or an alternative (sedentary video game or traditional active play).

SECONDARY OUTCOMES:
Change in minutes of physical activity, as assessed by activity tracker | Week 0, Week 6, Week 10
  Minutes of physical activity will be assessed by having participants wear an Actigraph accelerometer for 7 days (minimum 10 hours per day) on the right hip.
Change in minutes spent in traditional active play, active and sedentary video game play, and other sedentary screen-based activities | Week 0, Week 6, Week 10
  Changes in minutes spent in traditional active play, active and sedentary video game play, and other sedentary screen-based activities (computer, phone TV), will be assessed by 24-hour activity recalls which participants will fill out for the prior day's activities for two weekend and two weekdays.
Beverage and snack food consumption | Week 0, Week 6, Week 10
  Average weekly intake of certain foods and beverages will be assessed by self-report questionnaire responses of the Beverage and Snack Questionnaire (BSQ).
Children's exercise self-efficacy | Week 0, Week 6, Week 10
  Changes in children's exercise self-efficacy will be assessed by self-report questionnaire responses of the Children's Self-Perception of Adequacy in and Predilection of Physical Activity Scale (CSAPPA).
Children's intrinsic, external, interrogated, identified, introjected and amotivation for physical activity | Week 0, Week 6, Week 10
  Changes in children's intrinsic, external, interrogated, identified, introjected and amotivation for physical activity will be assessed by self-report questionnaire responses of the Behavioral Regulation in Exercise, 2nd Edition (BREQ-2).
Children's intrinsic, external, interrogated, identified, introjected and amotivation for active video game play | Week 0, Week 6, Week 10
  Changes in children's intrinsic, external, interrogated, identified, introjected and amotivation for active video game play will be assessed by self-report questionnaire responses of the Behavioral Regulation in Exercise, 2nd Edition (BREQ-2), modified to measure active video game play.
Children's intrinsic, external, interrogated, identified, introjected and amotivation for sedentary video game play | Week 0, Week 6, Week 10
  Changes in children's intrinsic, external, interrogated, identified, introjected and amotivation for sedentary video game play will be assessed by self-report questionnaire responses of the Behavioral Regulation in Exercise, 2nd Edition (BREQ-2), modified to measure sedentary video game play.

CONTACTS AND LOCATIONS:
Overall Officials: James N Roemmich, PhD, Principal Investigator — USDA Grand Forks Human Nutrition Research Center
Locations (1):
- USDA Grand Forks Human Nutrition Research Center, Grand Forks, North Dakota, United States

IPD SHARING:
Plan to Share IPD: No